CLINICAL TRIAL: NCT01753921
Title: Evaluation of a Non-invasive Brain Compliance Measurement Device
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Jan Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Tandy Aye, Assistant Professor, Stanford University
Other Study IDs: 22727
Record Dates: First submitted 2012-09-18; First posted 2012-12-20 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Diabetes; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DKA Group: Subjects who presented in diabetic ketoacidosis.
  Interventions: Other: this is not an intervention study; Device: MRI
- Healthy control: Control subjects without diabetes.
  Interventions: Other: this is not an intervention study; Device: MRI

INTERVENTIONS:
Other: this is not an intervention study — Subjects will wear the headband/helmet-like device for approximately 10 minutes on four different occasions: t=0, t=1week, t=1month, t=3months. Of note, part of the device also involves electrodes that are worn to obtain an electrocardiogram or EKG.
Other: this is not an intervention study — Subjects will be asked to participate in both computerized and non-computerized tests to assess subjects' cognitive (learning, language and memory) abilities, developmental level, and behavior. Tests will take place at t=0, t=1week, t=1month, t=3months.
Device: MRI — MRI study of the brain will be performed at t=3months.

SUMMARY:
This is a research study to understand how diabetic ketoacidosis may affect the brain and learning and to see if these changes are transient or permanent. The investigators hope to learn more about how diabetic ketoacidosis may cause changes in brain compliance (by wearing a non-invasive head band/helmet like device from Jan Medical: The Nautilus Neurowave System™ (NNS), learning, talking, behavior, or development. The investigators will compare those results from those with diabetes mellitus to those age and gendered matched healthy controls. Possible subjects in this study have diabetes mellitus and are between the ages of 10 to less than 17 years old OR do NOT have diabetes and are between the ages of 10 to less than 17 years old.

DETAILED DESCRIPTION:
At enrollment, 1 week, 1 month, 3 month, 12 month Computerized neurocognitive testing Wear NNS

MRI of the brain at 3 month and 12 months

Formal neurocognitive testing at 3 months and 12 months

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, all subjects must meet the following criteria:

1. Healthy control OR
2. Clinical new onset or established diagnosis of diabetes with diabetes ketoacidosis as defined by the Pediatric Endocrine Society Consensus Statement guidelines
3. Age 10 years to less than 17 years
4. Parent/guardian understand the study protocol and agrees to comply with it.
5. Primary care giver (i.e parent/guardian) comprehends written English. This is due to the fact that questionnaires and neurocognitive testing tools used as outcome measures do not have validated versions in Spanish or other language. Subject comprehends and speaks English.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for the study:

1. History of head trauma with any loss of consciousness
2. History of premature birth (less than 30 weeks of gestation)
3. History of significant developmental delay (lack of single word speech or ability to walk independently by 18 months of age
4. History of neurologic disease independent of diabetes (seizure disorder)

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 10-16 with DKA
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Unique signal measured in Hertz | 3 months
  We will be using the brain compliance measurement device to see if there is a unique signal for those with DKA and if so, follow the duration of this signal.

CONTACTS AND LOCATIONS:
Overall Officials: Tandy Aye, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- See also: Related Info — http://dped.stanford.edu/research/